CLINICAL TRIAL: NCT01248572
Title: Evaluation of Lens Effective Position, Stability and Prediction With a 12mm Uniplanar, Biaspheric Intraocular Lens
Brief Title: Evaluation of Effective Lens Position With a Uniplanar Bi-aspheric IOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lenstec Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LTHD-10-03
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Cataract
Keywords: Cataract; Biaspheric intraocular lens; Uniplanar intraocular lens; Effective lens position
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Softec HD IOL (Experimental)
  Interventions: Device: Softec HD IOL

INTERVENTIONS:
Device: Softec HD IOL — Posterior chamber intraocular lens intended for the replacement of the human crystalline lens following phacoemulsification cataract removal in adults over the age of 21.

SUMMARY:
The primary goal of this study is to determine the effective lens position (ELP) - or location an intraocular lens (IOL) "sits" in the eye - of the Softec HD IOL. A secondary study goal is to determine if measures of the eye taken prior to surgery can reliably predict postoperative ELP.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effective lens position (ELP) of the study lens, and to report the stability of ELP post-operatively. Additionally, correlations of ELP to predicted postoperative lens position, capsular bag metrics, preoperative biometry and age will be statistically analyzed for determination of ELP prediction via one, or a combination of preoperative variables.

ELIGIBILITY:
Inclusion Criteria:

* >=40 years of age, of any race and either gender
* Operable, age related cataract grade 3+ or lower in the study eye
* Able to achieve best corrected visual acuity (BCVA) 20/30 Snellen or better postoperatively in the study eye
* ≤1.0 diopter (D) of corneal astigmatism preoperatively in the study eye
* Able to achieve a dilated pupil >6.0 millimeter (mm) in the study eye
* Able to adequately visualize the lens equatorial diameter on ultrasound biomicroscopy (UBM) unit (preoperatively)
* Desire implantation of a monofocal lenses targeted at emmetropia in the study eye
* In good general and ocular health
* Able to competently complete testing
* Willing and able to attend study visits
* Willing and able to understand and sign an informed consent

Exclusion Criteria:

* Previous intraocular surgery or laser treatment
* Severe dry eye
* Uncontrolled IOP or glaucoma
* Retinal or macular pathology (i.e. macular degeneration, proliferative diabetic retinopathy, etc.)
* History of retinal detachment
* Microphthalmia
* Chronic severe uveitis
* Corneal decompensation
* Irregular astigmatism
* History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.)
* Clinically significant corneal endothelial dystrophy (e.g., Fuchs' dystrophy)
* Pseudoexfoliation syndrome
* Iris atrophy
* Pupil abnormalities (e.g., corectopia)
* Aniseikonia
* Amblyopia
* An acute or chronic disease or illness that may confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness)
* Pregnant, lactating, or planning to become pregnant during the course of the trial
* Participation in another clinical trial within 30 days of study start

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Effective Lens Position | 6 Months Postoperative
  The position of the intraocular lens - defined by measurement of the aqueous-containing space between the corneal endothelium and the anterior surface of the intraocular lens - once implanted in the capsular bag.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Barnet-Dulaney-Perkins Eye Center, Phoenix, Arizona
  - Eye Centers of Florida, Fort Myers, Florida
  - Harbin Clinic, Rome, Georgia